CLINICAL TRIAL: NCT06947499
Title: A Prospective, Multi-national, Multi-center, Open-label, Randomized, Active Controlled, Parallel Group, Operationally Seamless Phase II/III Clinical Study to Evaluate the Immunogenicity, Safety and Lot-to-lot Consistency of LBVD, a Fully Liquid Hexavalent Diphtheria-tetanus-whole Cell Pertussis-hepatitis B-poliovirus (Inactivated)-Haemophilus Influenzae Type b Conjugate (DTwP-HepB-IPV-Hib) Vaccine, Compared to Co-administration of DTwP-HepB-Hib Vaccine and IPV Vaccine in Healthy Infants at 6-, 10-, and 14-week of Age as Primary Series
Brief Title: A Phase II/III Study to Evaluate the Immunogenicity, Safety and Lot-to-lot Consistency of LBVD, a Fully Liquid Hexavalent Diphtheria-tetanus-whole Cell Pertussis-hepatitis B-poliovirus-Haemophilus Influenzae Type b Conjugate (DTwP-HepB-IPV-Hib) Vaccine, in Healthy Infants as Primary Series
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VDCL004
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type b
Keywords: vaccination
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — Vaccines, Combined; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Test group 1 for Stage 1 (Experimental): LBVD
  Interventions: Biological: LBVD
- Test group 1 for Stage 2 (Experimental): LBVD Lot A
  Interventions: Biological: LBVD
- Test group 2 for Stage 2 (Experimental): LBVD Lot B
  Interventions: Biological: LBVD
- Test group 3 for Stage 2 (Experimental): LBVD Lot C
  Interventions: Biological: LBVD
- Control group for Stage 1 and Stage 2 (Active Comparator): Co-administration of Pentavalent vaccine and Inactivated Polio vaccine
  Interventions: Biological: Pentavalent vaccine and Inactivated Polio vaccine

INTERVENTIONS:
Biological: LBVD — Intramuscular injection into the anterolateral area of the thigh
  Arms: Test group 1 for Stage 1; Test group 1 for Stage 2; Test group 2 for Stage 2; Test group 3 for Stage 2
Biological: Pentavalent vaccine and Inactivated Polio vaccine — Intramuscular injection into the anterolateral area of the thigh
  Arms: Control group for Stage 1 and Stage 2

SUMMARY:
The purpose of this study is to evaluate immunogenicity, safety and lot-to-lot consistency of LBVD in comparison to co-administration of Pentavalent vaccine and Poliomyelitis Vaccine (Inactivated) in separate injections at four weeks after completion of three-dose primary series at 6-10-14 weeks of age when administered to healthy infants

DETAILED DESCRIPTION:
Stage 1 (Phase 2)

1. To compare the immunogenicity and safety of LBVD to the licensed Control vaccines at 4 weeks after a three-dose primary series of vaccination given at 6-, 10- and 14-week of age

Stage 2 (Phase 3)

1. To demonstrate the non-inferior immunogenicity of LBVD to the licensed Control Vaccine at 4 weeks after a three-dose primary series of vaccination given at 6-, 10- and 14-week of age
2. To demonstrate lot-to-lot consistency in the immunogenicity of three separate lots of LBVD at 4 weeks after a three-dose primary series of vaccination given at 6-, 10- and 14-week of age

ELIGIBILITY:
Inclusion Criteria:

* healthy infants from 6 weeks to 8 weeks of age (both inclusive)
* body weight ≥ 3.2 kg
* born at full term pregnancy (≥ 37 weeks)
* signed informed consent by parent(s) or legally acceptable representative(s)

Exclusion Criteria:

* Known history of Hib infection, HepB, diphtheria, tetanus, pertussis, or poliomyelitis
* Household contact or intimate exposure with a confirmed case of Hib, HepB, diphtheria, pertussis, tetanus or poliomyelitis within 30 days prior to study registration
* Known history of SARS-CoV-2 infection
* Participant's mother is HepB antigen or HIV positive
* Fever ≥ 38.0 C/100.4 F within 3 days prior to enrollment
* Vaccination history of non-study vaccines within 30 days prior to enrollment except for pneumococcal conjugate, rotavirus, HepB and Bacillus Calmette Guerin (BCG)
* Previous use of any diphtheria, tetanus, pertussis-based combination vaccine(s), Hib conjugate, poliovirus, or combination
* Received immunosuppressive agents or other immune-modifying drugs
* Previous use of blood or blood-derived products
* Any history of allergy (hypersensitivity) to any of the vaccine components
* Participation in another interventional clinical trial within 4 weeks of expected first vaccination

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1186 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Seroprotection/seroconversion rate | 4 weeks after a three-dose primary series
  proportion of participants achieving pre-defined immune response to each antigen
Geometric mean concentration (GMC) for pertussis | 4 weeks after a three-dose primary series
  GMC for pertussis antigen

SECONDARY OUTCOMES:
Geometric mean titer (GMT) or GMC | 4 weeks after the three-dose primary series
  GMT or GMC for all antigens
Seroprotection/seroconversion rate | 4 weeks after the three-dose primary series
  Proportion of participant achieving pre-defined immune response to each antigen
Immediate reactions after vaccination | 30 minutes after each vaccination
  any signs and symptoms which occur within the first 30 minutes after each vaccination will be monitored
Solicited adverse event | within 7 days after each vaccination
  local or systemic signs and symptoms
Unsolicited adverse event | 4 weeks after the three-dose primary series
  All adverse events other than solicited adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Care CT Group, Dasmariñas, Cavite, Philippines